CLINICAL TRIAL: NCT01129778
Title: Assessment of the Effects of Zegerid Powder for Oral Suspension 40 mg on 24-Hour and Nocturnal Esophageal Acid Exposure in Patients With Gastroesophageal Reflux Disease and Barrett's Esophagus
Brief Title: Assessment of Zegerid on Esophageal pH in Patients With Barrett's Esophagus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: change in the business strategy of the sponsor
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-04302010-5803
Record Dates: First submitted 2010-05-21; First posted 2010-05-25 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Barrett Esophagus; Gastroesophageal Reflux
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux | interventions — omeprazole, sodium bicarbonate drug combination; Proton Pump Inhibitors

ARMS (1):
- Received Zegerid (Ome-NaBic) (Experimental): Administered Ome-NaBic 40 mg orally 1 h before breakfast and bedtime
  Interventions: Drug: Zegerid (proton pump inhibitor); Procedure: Bravo pH monitoring

INTERVENTIONS:
Drug: Zegerid (proton pump inhibitor)
  Other Names: Omeprazole-sodium bicarbonate (Ome-NaBic)
Procedure: Bravo pH monitoring

SUMMARY:
The purpose of this research study is to assess how safe, effective (how well it works), and tolerable (to put up with) the drug Zegerid is in reducing reflux episodes in patients who have both gastroesophageal reflux disease (GERD) and Barrett's esophagus. Zegerid has been approved by the US Food and Drug Administration (FDA) for the treatment of GERD. The investigators hope to learn the effectiveness of Zegerid for reducing the amount of acid reflux patients are experiencing in the esophagus (swallowing pipe).

DETAILED DESCRIPTION:
The following procedures will be performed at the Screening Visit:

* Obtain informed consent.
* Obtain information about your age and gender.
* Evaluate whether you qualify for the study.
* Document prior negative testing for H. pylori infection (a bacterial infection in the stomach that can cause ulcers) including the date of testing.
* Make sure that you have not used any investigational medications or participated in a clinical trial in the 30 days prior to the Screening Visit.
* Obtain medical history.
* Record medication history (including concomitant medications).
* Obtain vital signs.
* Conduct a physical examination.
* If a Bravo pH study has not been done within 8 weeks, instruct the patient to discontinue their medication for GERD during the 7-10 day washout period.
* Instruct the patient to discontinue the use of all prohibited medications during the applicable time intervals and not to start any new concomitant medications during the trial.
* Distribute Gelusil tablets to be used as "rescue medication"; instruct the patient that no more than 6 Gelusil tablets per day or 21 tablets over any 7-day interval will be allowed.
* Schedule the patient to return for the Qualification Visit, or for pH monitoring and the Qualification Visit. Only patients with abnormal pH monitoring will be able to enter the treatment period.

Procedures that will occur during the Treatment Period:

* You will receive Zegerid 1 hour before breakfast and at bedtime for at least 14 days and no longer than 28 days
* At the end of the Zegerid treatment period, you will undergo 48-hour Bravo pH monitoring on Zegerid therapy for two days. You will complete a symptom survey and quality of life survey after the completion of the pH study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include adult men and women (aged <=18 years) with previously established, biopsy-proven diagnosis of BE (any length intestinal metaplasia without dysplasia or adenocarcinoma)

Exclusion Criteria:

* Exclusion criteria include a history of esophageal, gastric, or duodenal surgery (including antireflux surgery or endoscopic antireflux procedures), except for simple ulcer closure
* Zollinger-Ellison syndrome
* Endoscopic evidence or suspicion of a pathologic or infiltrative process in the stomach
* Positive for H. pylori.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren B Gerson, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- See also: Link to publication about this study — http://onlinelibrary.wiley.com/doi/10.1111/j.1365-2036.2012.05016.x/full

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants withdrew after providing their informed consent and before beginning their participation in the study.
Groups:
- Received Zegerid (Ome-NaBic): Ome-NaBic 40 mg orally 1 h before breakfast and bedtime for up to 29 days
Period: Overall Study
Arm/Group | Received Zegerid (Ome-NaBic)
Started | 22
Completed | 15
Not Completed | 7

BASELINE CHARACTERISTICS:
Population: 21 participants who underwent pH testing were evaluable for Baseline Characteristics.
Arm/Group | Received Zegerid (Ome-NaBic)
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 17
Mean RDQ heartburn score [Mean (Standard Deviation); unit: units on a scale] — The RDQ is a 12 item survey that asks the patient to rate the frequency and severity of GERD symptoms. Each item is scored from 0 to 5 where a score of 0 is equivalent to an asymptomatic state and 5 indicates the worst severity of GERD symptoms. The total RDQ is a sum of all 12 items, and can range from 0 to 60.
  units on a scale | 10 (6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time Esophageal pH< 4
Description: Reported as the the average percentage over 24 hours of total time, upright time, and supine time per day with pH <4 (symptomatic acid state) as evaluated with the Bravo pH monitoring technique.
Time Frame: Days 1 and 2
Population: Participants who completed all protocol-specified assessments were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of hours
Arm/Group | Received Zegerid (Ome-NaBic)
Number analyzed (Participants) | 15
percentage of hours
  Total time pH <4 First Day | 0.4 (0.5)
  Total time pH <4 Second Day | 0.6 (1.8)
  Upright time pH <4 First Day | 0.7 (0.7)
  Upright time pH <4 Second Day | 1 (3)
  Supine time pH <4 First Day | 0.06 (0.1)
  Supine time pH <4 Second Day | 0.05 (0.2)

2. Secondary Outcome: Reflux Disease Questionnaire Score on Day 1 After Therapy Completion
Description: The RDQ is a 12 item survey that asks the patient to rate the frequency and severity of GERD symptoms. Each item is scored from 0 to 5 where a score of 0 is equivalent to an asymptomatic state and 5 indicates the worst severity of GERD symptoms. The total RDQ is a sum of all 12 items, and can range from 0 to 60.
Time Frame: Day 1 after therapy period completion
Population: Participants who completed all protocol-specified assessments were included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Received Zegerid (Ome-NaBic)
Number analyzed (Participants) | 15
Units on a scale | 0.5 (1.5)

ADVERSE EVENTS:
Arm/Group | Received Zegerid (Ome-NaBic)
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

LIMITATIONS AND CAVEATS:
The limitations included the small sample size, a cohort of patients with primarily short-segment BE, and the fact that the study relied on comparison of intraoesophageal pH levels on Ome-NaBic to other PPIs based on historical controls.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes